CLINICAL TRIAL: NCT03236129
Title: Allogeneic Immunotherapy for Hematological Malignancies by Selective Depletion of Regulatory T Cells: A Confirmatory, Randomized, Double Blinded Trial
Brief Title: Allogeneic Immunotherapy for Hematological Malignancies by Selective Depletion of Regulatory T Cells
Acronym: DLI-Boost
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P140303; 2016-A00645-46 (Other: IDRCB)
Record Dates: First submitted 2017-07-05; First posted 2017-08-01 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Hematological Malignancies; Regulatory T Cell Depletion; Relapse
Keywords: DLI; Regulatory T cells depletion; Hematological malignancies; Relapse
MeSH Terms: conditions — Hematologic Neoplasms; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treg depleted DLI (Experimental): Patients will receive a lymphodepleting treatment combining cyclophosphamide and fludarabine followed by Treg depleted (Donor Lymphocytes Infusion (DLI)
  Interventions: Procedure: T-reg depleted DLI
- Unmanipulated DLI (Active Comparator): Patients will receive a lymphodepleting treatment combining cyclophosphamide and fludarabine followed by a standard DLI (unmanipulated)
  Interventions: Procedure: Standard DLI

INTERVENTIONS:
Procedure: T-reg depleted DLI — The patients in the experimental arm benefit of a DLI depleted from regulatory T lymphocytes
  Arms: Treg depleted DLI
Procedure: Standard DLI — The patients in this arm benefit of a standard DLI.
  Arms: Unmanipulated DLI

SUMMARY:
The investigators have previously shown the absence of toxicity of Treg-depleted-DLI and the possibility to triggering alloreactivity (GVHD/GVT) in relapsing patients dealing with hematological malignancies who had never shown any signs of GVHD after transplant or after one or more DLI.

The Investigators, we plan to demonstrate the benefit of Treg-depleted DLI as compared to the reference treatment of relapse in hematological malignancies after allogeneic HSCT which is currently based on standard DLI

DETAILED DESCRIPTION:
This clinical trial is designed to demonstrate the benefit of Treg-depleted DLI as compared to the reference treatment of relapse in hematological malignancies after allogeneic HSCT which is currently based on standard DLI.

Patients who have never shown any signs of GVHD and for which one (or more) unmanipulated DLI have been ineffective. Those patients will receive a subsequent DLI, which will be either unmanipulated (control arm) or Treg depleted (experimental arm) after a randomization. In both cases, the second DLI will be immediately preceded by a lymphodepleting treatment based on cyclophosphamide and fludarabine association.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults regardless of age or weight allograft for primary or secondary acute leukemia, MDS, lympho-proliferative syndrome (CLL, Myeloma, Lymphoma) or myelo-proliferative syndrome.
* Prior allogeneic HSCT (myeloablative or non-myeloablative conditioning) from a family donor geno-identical HLA or a volunteer donor HLA 10/10 or 9/10.
* Molecular, cytogenetic, cytological relapse regardless of the date after the transplant.
* Previous standard DLI should have brought a total dose of at least 5.10^6 CD3 + / kg (donor HLA-geno idendique) or 2.10^6 CD3 + / kg (voluntary donor) or 5.10^5 CD3+/kg (donor haplo-idendique).
* Patient corresponding to the failure criteria of a previous standard DLI, defined for each type of hematological malignancies in the test model "DLI-Treg-1" after a delay of at least 30 days in the case of a progressive disease after DLI and at least 60 days in the case of stable disease (due to possible delayed responses after DLI).
* Patient consented to the study (the consent of both parents will be collected for minors)
* Patients insured by a social security system.
* Negative pregnancy test (β-HCG hormone) within the 7 days prior to enrollment

Exclusion Criteria:

* Presence of acute GVHD grade> II or extensive chronic GVHD since the first DLI
* Patient receiving immunosuppressive therapy for the treatment of GVHD or other reason
* Impairment of liver function (transaminases> 5 N or bilirubin> 50 µM except Gilbert's disease) or renal function (creatinine clearance <30 ml / min)
* OMS performance status > 2
* Non controlled severe infection
* Patient under tutorship, curatorship or legal protection

Donor Inclusion Criteria

* Being the initial HSC donor (HLA geno-identical family or haplo-identique or non-family HLA 10/10 or 9/10)
* Weight ≥20 kg authorizing the lymphapheresis
* Having no contra-indications for donating blood
* Absence of severe heart failure, unstable heart disease, uncontrolled hypertension, type 1 diabetes
* Negative serology for HIV1-2, HBV, HCV, HTLV 1 and VDRL/TPHA in the 30 days prior to apheresis. Negative viral genomics diagnosis is required for HIV, HBV and HCV
* Being informed of the study, and have given an oral non opposition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of clinical manifestations of GVHD, in the form of acute GVHD with grade ≥ 2 and/or extensive chronic. This parameter will take into account the competitive risk of death unrelated to the GVHD | 3 month after injection

SECONDARY OUTCOMES:
Cumulative incidence of relapse, taking into account the competitive risk of death unrelated to relapse | 1 year after injection
Relapse-free survival | 1 year after injection
Overall survival | 1 year after injection

CONTACTS AND LOCATIONS:
Overall Officials: Florence BEKCERICH, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maury S, Lemoine FM, Hicheri Y, Rosenzwajg M, Badoual C, Cherai M, Beaumont JL, Azar N, Dhedin N, Sirvent A, Buzyn A, Rubio MT, Vigouroux S, Montagne O, Bories D, Roudot-Thoraval F, Vernant JP, Cordonnier C, Klatzmann D, Cohen JL. CD4+CD25+ regulatory T cell depletion improves the graft-versus-tumor effect of donor lymphocytes after allogeneic hematopoietic stem cell transplantation. Sci Transl Med. 2010 Jul 21;2(41):41ra52. doi: 10.1126/scitranslmed.3001302. PMID 20650872